CLINICAL TRIAL: NCT06505551
Title: A Phase 1/2 Open Label, Single Arm, Multicenter Study to Evaluate the Safety and Preliminary Eficacy of Autologous SCG142 T Cell Receptor (TCR) T Cells in Patients With Advanced or Metastatic HPV16- or HPV52-positive Carcinomas
Brief Title: Phase 1/2 Study of Autologous SCG142 TCR T Cells in Patients With HPV16/52-positive Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCG Cell Therapy Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCG142-UR-102
Record Dates: First submitted 2024-07-01; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: HPV-Related Squamous Cell Carcinoma; HPV-Related Cervical Squamous Cell Carcinoma; HPV-Related Vulvar Squamous Cell Carcinoma; HPV-Related Penile Squamous Cell Carcinoma; HPV-Related Vaginal Squamous Cell Carcinoma; HPV-Related Anal Squamous Cell Carcinoma; HPV-Related Head and Neck Cancer
Keywords: Human Papilloma Virus; HPV; Cervical Cancer; Head and Neck Cancer; Oropharyngeal Cancer; Vulvar Cancer; Vaginal Cancer; Penile Cancer; Anal Cancer; Anogenital Cancer; TCR T Cell; Cell therapy; T cell receptor T cell
MeSH Terms: conditions — Head and Neck Neoplasms; Uterine Cervical Neoplasms; Oropharyngeal Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Penile Neoplasms; Anus Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SCG142 T cells (Experimental): This is a single arm study.
  Interventions: Biological: SCG142; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: SCG142 — Autologous SCG142 cells infused on Day 0 after completion of lymphedepletion chemotherapy
Drug: Cyclophosphamide — for 3 consecutive days
Drug: Fludarabine — for 3 consecutive days

SUMMARY:
This is a phase 1/2, open-label, single arm, multicenter study in patients with advanced or metastatic HPV16- or HPV52-positive carcinomas who have progressed after at least one line of systemic therapy, including but not limited to combination chemotherapy and/or combination chemo-immunotherapy

DETAILED DESCRIPTION:
This study will be conducted in 2 parts:

The Phase 1 part of the trial consists of a dose-escalation portion designed to evaluate the safety and tolerability of SCG142, and to identify the RP2D.

The Phase 2 part of the trial is designed to evaluate the preliminary efficacy of SCG142 in the same patient populations.

ELIGIBILITY:
Main Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma (SCC); may include any of the following tumor types: cervical, head and neck, anal, penile, vulvar, or vaginal.
2. Tumor tissue positive for HPV16 or HPV52.
3. Advanced or metastatic carcinoma with progression after at least 1 line of standard of care systemic therapies, including but not limited to combination chemotherapy and/or combination chemo-immunotherapy.
4. Human leukocyte antigen (HLA)-A*02:01 genotype.
5. Measurable disease as defined by RECIST v1.1.
6. Eastern Cooperative Group (ECOG) Performance Status of 0 or 1.
7. Anticipated life expectancy ≥3 months.
8. Adequate laboratory parameters including hematologic, renal, hepatic and coagulation function.

Main Exclusion Criteria:

1. Presence of clinically relevant or active seizure disorder, stroke, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with central nervous system (CNS) involvement.
2. Active brain metastasis or leptomeningeal metastases.
3. History of other malignancy within 2 years prior to Screening.
4. History of organ transplant.
5. Positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
6. History of active cardiac disease.
7. History of active pulmonary disease.
8. Active, known, or suspected autoimmune disease.
9. Lack of peripheral venous or central venous access, or any condition that may prevent trial sample collection and administration of SCG142.
10. Prior exposure to any cell therapy including, but not limited to natural killer (NK) cells, cytokine-induced killer (CIK) cells, dendritic cells (DCs), cytotoxic T lymphocytes (CTLs), stem cell therapy, and CAR/TCR-T cell therapy.
11. Allergy to LD chemotherapy (cyclophosphamide or fludarabine) and/or any component of SCG142.
12. Any serious medical condition or abnormality in clinical laboratory tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Phase 1) | 2 years
  Incidence of dose-limiting toxicities (DLTs) and occurrence of study related adverse events.
Objective response rate (ORR) (Phase 2) | 2 years
  The proportion of patients with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Objective response rate (ORR) (Phase 1) | 2 year
  The proportion of patients with a complete response (CR) or partial response (PR)
Duration of objective response (DOR) (Phase 1&2) | 2 year
  The time from the first occurrence of a confirmed response to disease progression or death from any cause
Disease control rate (DCR) (Phase 1&2) | 2 year
  The proportion of patients with a CR, PR or stable disease (SD)
Progression-free survival (PFS) (Phase 1&2) | 2 year
  The time from the date of the SCG142 administration to the first occurrence of a progressive disease (PD) or death from any cause
Overall survival (OS) (Phase 1&2) | 2 year
  The time from date of the SCG142 administration to date of death of any cause
Incidence of Treatment-Emergent Adverse Events (Phase 2) | 2 years
  TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: SCG Cell Therapy, Study Director — SCG Cell Therapy Pte. Ltd.

IPD SHARING:
Plan to Share IPD: No